CLINICAL TRIAL: NCT05463679
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study of Enzastaurin for the Prevention of Arterial Events in Patients With Vascular Ehlers-Danlos Syndrome (vEDS) Confirmed With COL3A1 Mutations, Followed by an Open Label Extension (OLE)
Brief Title: Investigate Efficacy, Safety, and Pharmacokinetics of Enzastaurin for the Prevention of Arterial Events in Patients With Vascular Ehlers-Danlos Syndrome.
Acronym: PREVEnt
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Indefinite hold by company
Sponsor: Aytu BioPharma, Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AR101-PREVEnt
Record Dates: First submitted 2022-04-06; First posted 2022-07-19 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Vascular Ehlers-Danlos Syndrome
MeSH Terms: conditions — Ehlers-Danlos Syndrome, Type IV | interventions — enzastaurin

STUDY DESIGN:
Intervention Model Description: Two-arm, multicenter, randomized, double-blind, placebo-controlled study in patients with vEDS receiving enzastaurin 500 mg once daily (QD) compared to placebo, in addition to background standard of care, followed by an OLE phase.
  Approximately 260 patients with vEDS are planned to be randomized in a 1:1 ratio of enzastaurin or placebo. Patients will be enrolled in the study if they meet all eligibility criteria.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enzastaurin 500 mg QD (Active Comparator): Receive 500 mg enzastaurin QD plus background standard of care.
  Interventions: Drug: Enzastaurin
- Placebo QD (Placebo Comparator): Matching placebo QD plus background standard of care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enzastaurin — 500 mg QD orally in the form of four 125 mg tablets with background standard of care
  Arms: Enzastaurin 500 mg QD
Drug: Placebo — Placebo to match enzastaurin 500 mg QD orally in the form of four 125 mg tablets with background standard of care
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to investigate the efficacy of enzastaurin compared to placebo in preventing arterial events (rupture, dissection, pseudoaneurysm, carotid-cavernous sinus fistula, or aneurysm, fatal or not) leading to intervention or mortality attributable to an arterial event in patients with vEDS confirmed with pathogenic heterozygous COL3A1 gene mutations predicted to derive a mutant protein.

DETAILED DESCRIPTION:
The primary efficacy endpoint of this study will be defined as the time to intervention for an arterial event (rupture, dissection, pseudoaneurysm, carotid-cavernous sinus fistula, or aneurysm, fatal or not) or mortality attributable to an arterial event, as adjudicated by an Event Committee, and will be analyzed for difference of active vs. placebo treatments on top of background standard of care, using survival statistical analysis. Furthermore, secondary endpoints will include the rate of intestinal rupture, pneumothorax, and retinal detachment, as adjudicated by an Event Committee, safety and tolerability, as well as hospitalizations and Health Related Quality of Life (HQRL) measures.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 - 60 years old at time of initial screening.
2. Adolescent subjects aged 12 - 17 years old, may be considered to enroll later in the clinical trial pending interim analysis.
3. Diagnosis for VEDS (vascular Ehlers Danlos Syndrome), with a confirmed and documented COL3A1 genetic variant.
4. Subject should be stable, having no VEDS-related vascular events within the past 3 months prior to enrollment.
5. Confirmed use of contraception for both male and female participants.

Exclusion Criteria:

1. Inability to swallow or receive intact tablets.
2. Currently being treated with CYP3A4 inhibitors within 4 weeks prior to enrollment.
3. Known allergy or hypersensitivity to enzastaurin.
4. Patient currently pregnant or breast feeding.

Other criteria will be reviewed at the first study visit to determine if you are able to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Time to intervention for an arterial event (rupture, dissection, pseudoaneurysm, carotid-cavernous sinus fistula, or aneurysm, fatal or not) or mortality attributable to an arterial event. | 30 months
  Time to intervention for an arterial event (rupture, dissection, pseudoaneurysm, carotid-cavernous sinus fistula, or aneurysm, fatal or not) or mortality attributable to an arterial event, as adjudicated by an Event Committee and analyzed for difference in the time-to-composite-event of active vs. placebo treatments, using survival analysis until end of study

SECONDARY OUTCOMES:
Number of and proportion of patients with adverse events, or with abnormal vital signs, physical examinations, ophthalmological examinations, clinical laboratory values, or electrocardiograms (ECGs) medical attention. | 30 months
  An Adverse Event (AE) is defined as any untoward medical occurrence associated with the use of the investigational product in humans, whether or not considered related to investigational product. An AE can be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with any use of the investigational product, without any judgment about causality and irrespective of route of administration, formulation, or dose, including an overdose.
Number of and proportion of patients who discontinue study drug due to adverse events | 30 months
  Discontinuation or withdrawal from the study

CONTACTS AND LOCATIONS:
Overall Officials: Sherene Shalhub, M.D., M.P.H., Principal Investigator — University of Washington; Shaine Morris, M.D.,M.P.H., Principal Investigator — Texas Children's Hospital and Baylor College of Medicine
Locations (1):
- Aytu BioPharma, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowen CJ, Calderon Giadrosic JF, Burger Z, Rykiel G, Davis EC, Helmers MR, Benke K, Gallo MacFarlane E, Dietz HC. Targetable cellular signaling events mediate vascular pathology in vascular Ehlers-Danlos syndrome. J Clin Invest. 2020 Feb 3;130(2):686-698. doi: 10.1172/JCI130730. PMID 31639107
- See also: 2. Bowen CJ et al. Targetable cellular signaling events mediate vascular pathology in vascular Ehlers-Danlos Syndrome. J Clin Invest. 2020 Feb 3;130(2):686-698. — https://www.clinicaltrials.gov/ct2/show/NCT00332202